CLINICAL TRIAL: NCT06121973
Title: The Effects of Video-Assisted Breastfeeding Education Given to Primiparous Pregnant Women on Breastfeeding Self-Efficacy: Randomised Control Study
Brief Title: The Effects of Video-Assisted Breastfeeding Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ayşe Metin, Assist. Prof., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 7412169
Record Dates: First submitted 2023-10-27; First posted 2023-11-08 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Related; Breastfeeding; Breastfeeding, Exclusive; Educational Problems
Keywords: Pregnancy; Breastfeeding self-efficacy; Breastfeeding education; Video-assisted education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Pregnant women in the control group did not receive any intervention other than routine care.
- Experimental group (Experimental): Pregnant women in the intervention group received online video-assisted education which demonstrated first meeting of the mother-baby and first breastfeeding in addition to receiving counselling on breastfeeding.
  Interventions: Behavioral: educational group

INTERVENTIONS:
Behavioral: educational group — Experimental group received online video-supported breastfeeding education in an online classroom for 6-8 people and individual counselling via phone and Whatsapp application when needed for 3 weeks.
  Arms: Experimental group

SUMMARY:
The present study was conducted to determine the effects of online video-assisted breastfeeding education on breastfeeding self-efficacy in primiparous pregnant women.

DETAILED DESCRIPTION:
This two-group parallel randomized controlled study was conducted with pregnant women admitted to the pregnancy follow-up outpatient clinics of a university hospital in northern Turkey. The study was completed with 80 pregnant women in their second trimester, 40 pregnant women each in the intervention and control groups. Pregnant women in the intervention group received online video-assisted education which demonstrated first meeting of the mother-baby and first breastfeeding in addition to receiving counselling on breastfeeding. Pregnant women in the control group did not receive any intervention other than routine care. Data were collected face-to-face with the breastfeeding self-efficacy scale at the beginning of the study and two weeks later. In data analysis, chi-square test was used for categorical variables, independent sample t-test was used for continuous variables and intergroup comparison, and paired sample t-test was used for intragroup comparison.

ELIGIBILITY:
Inclusion Criteria:

* Having a primiparous pregnancy
* Pregnant woman in the second trimester
* There is no risk during pregnancy
* Pregnant woman's ability to read and write
* Volunteering to participate in the study

Exclusion Criteria:

* Having auditory problems
* Having visual problems
* Having psychological problems
* Having cognitive problems
* Wanting to leave work

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Prenatal Breastfeeding Self-Efficacy Scale (PBSES) | 5 Minutes
  The scale was developed by Wells et al. (2006) to determine the breastfeeding self-efficacy perceptions of pregnant women in the prenatal period.(27) Turkish validity and reliability of the scale was conducted by Aydın and Pasinlioğlu (2016). The scale consists of a total of 20 items. Each item of the scale is a 5-point Likert scale ranging between "1=Not at all sure - 5= Completely sure". Minimum 20 and maximum 100 points can be obtained from the scale. Higher score indicates breastfeeding self-efficacy perception. Cronbach's alpha value of the scale was reported to be 0.86.(28) Cronbach's alpha value was found to be 0.96 in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Metin, Study Director — Erzurum Technical University
Locations (1):
- Ayşe Metin, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are not publicly available due to the sensitive nature of the interviews. If someone wants to request the data from this study, the corresponding author should be contacted.

REFERENCES:
- [Background] Yuen M, Hall OJ, Masters GA, Nephew BC, Carr C, Leung K, Griffen A, McIntyre L, Byatt N, Moore Simas TA. The Effects of Breastfeeding on Maternal Mental Health: A Systematic Review. J Womens Health (Larchmt). 2022 Jun;31(6):787-807. doi: 10.1089/jwh.2021.0504. Epub 2022 Apr 18. PMID 35442804
- [Background] Piro SS, Ahmed HM. Impacts of antenatal nursing interventions on mothers' breastfeeding self-efficacy: an experimental study. BMC Pregnancy Childbirth. 2020 Jan 6;20(1):19. doi: 10.1186/s12884-019-2701-0. PMID 31906881
- [Background] Karacam Z, Kitis Y. What do midwives and nurses in Turkey know about nutrition in the first six months of life. Midwifery. 2005 Mar;21(1):61-70. doi: 10.1016/j.midw.2004.09.005. PMID 15740817
- [Background] Perez-Escamilla R, Tomori C, Hernandez-Cordero S, Baker P, Barros AJD, Begin F, Chapman DJ, Grummer-Strawn LM, McCoy D, Menon P, Ribeiro Neves PA, Piwoz E, Rollins N, Victora CG, Richter L; 2023 Lancet Breastfeeding Series Group. Breastfeeding: crucially important, but increasingly challenged in a market-driven world. Lancet. 2023 Feb 11;401(10375):472-485. doi: 10.1016/S0140-6736(22)01932-8. Epub 2023 Feb 7. PMID 36764313
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Kartal T, Gursoy E. Sürdürülebilir Kalkınma Amaçlarında (2015-2030) Emzirmenin Önemi ve Türkiye'deki Mevcut Durum Işığında Hemşireye Düşen Görevler. Mersin Üniversitesi Tıp Fakültesi Lokman Hekim Tıp Tarihi ve Folklorik Tıp Dergisi. 2020;10(2):147-53. https://doi.org/10.31020/mutftd.676389
- [Background] Meek JY, Noble L; Section on Breastfeeding. Policy Statement: Breastfeeding and the Use of Human Milk. Pediatrics. 2022 Jul 1;150(1):e2022057988. doi: 10.1542/peds.2022-057988. PMID 35921640
- [Background] Wu Q, Tang N, Wacharasin C. Factors influencing exclusive breastfeeding for 6 months postpartum: A systematic review. Int J Nurs Knowl. 2022 Oct;33(4):290-303. doi: 10.1111/2047-3095.12360. Epub 2022 Jan 28. PMID 35088945
- [Background] McGovern L, Geraghty A, McAuliffe F, O'Reilly S. An exploration of prenatal breastfeeding self-efficacy: a scoping review protocol. Open Res Eur. 2023 Jan 24;2:91. doi: 10.12688/openreseurope.14938.3. eCollection 2022. PMID 37645344
- [Background] Dennis CL. Theoretical underpinnings of breastfeeding confidence: a self-efficacy framework. J Hum Lact. 1999 Sep;15(3):195-201. doi: 10.1177/089033449901500303. No abstract available. PMID 10578797
- [Background] Ummah F, Rosida L. Breastfeeding Self Efficacy Among Pregnant Women. Jurnal EduHealth. 2022;13(01):336-42.
- [Background] Ghasemi V, Simbar M, Banaei M, Saei Ghare Naz M, Jahani Z, Nazem H. The effect of interventions on breastfeeding self-efficacy by using Bandura's theory in Iranian mothers: a systematic review. International Journal of Pediatrics. 2019;7(8):9939-54. https://doi.org/10.22038/ijp.2019.40842.3446
- [Background] Ozturk R, Ergun S, Ozyazicioglu N. Effect of antenatal educational intervention on maternal breastfeeding self-efficacy and breastfeeding success: a quasi-experimental study. Rev Esc Enferm USP. 2022 Apr 4;56:e20210428. doi: 10.1590/1980-220X-REEUSP-2021-0428. eCollection 2022. PMID 35377385
- [Background] Demirci J, Caplan E, Murray N, Cohen S. "I Just Want to Do Everything Right:" Primiparous Women's Accounts of Early Breastfeeding via an App-Based Diary. J Pediatr Health Care. 2018 Mar-Apr;32(2):163-172. doi: 10.1016/j.pedhc.2017.09.010. Epub 2017 Dec 21. PMID 29276003
- [Background] Chantry CJ, Dewey KG, Peerson JM, Wagner EA, Nommsen-Rivers LA. In-hospital formula use increases early breastfeeding cessation among first-time mothers intending to exclusively breastfeed. J Pediatr. 2014 Jun;164(6):1339-45.e5. doi: 10.1016/j.jpeds.2013.12.035. Epub 2014 Feb 14. PMID 24529621
- [Background] Lopez EP, Gonzalez S, Sanchez M. Educational intervention for the main caregiver of primiparous women to promote breastfeeding and the association between prolactin and nutritional parameters. J Glob Health. 2023 Apr 21;13:04046. doi: 10.7189/jogh.13.04046. PMID 37083003
- [Background] Uzuncakmak T, Goksin I, Ayaz-Alkaya S. The effect of social media-based support on breastfeeding self-efficacy: a randomised controlled trial. Eur J Contracept Reprod Health Care. 2022 Apr;27(2):159-165. doi: 10.1080/13625187.2021.1946500. Epub 2021 Jul 12. PMID 34251949
- [Background] Littleton-Gibbs LY, Engebretson J. Maternity Nursing Care (Book Only): Cengage Learning; 2012.
- [Background] Yanıkkerem E, Ay S, Göker A. Primipar ve multipar gebelerin emzirme tutumu ve yaşadıkları endişeler. Van Tıp Dergisi. 2014;21(1):6-16.
- [Background] Taylor AM, Hutchings M. Using video narratives of women's lived experience of breastfeeding in midwifery education: exploring its impact on midwives' attitudes to breastfeeding. Matern Child Nutr. 2012 Jan;8(1):88-102. doi: 10.1111/j.1740-8709.2010.00258.x. Epub 2010 Aug 16. PMID 22136222
- [Background] Akyildiz D, Bay B. The effect of breastfeeding support provided by video call on postpartum anxiety, breastfeeding self-efficacy, and newborn outcomes: A randomized controlled study. Jpn J Nurs Sci. 2023 Jan;20(1):e12509. doi: 10.1111/jjns.12509. Epub 2022 Sep 7. PMID 36071624
- [Background] Sari Ozturk C, Demir K. The Effect of Mandala Activity and Technology-Based Breastfeeding Program on Breastfeeding Self-Efficacy and Mother-Infant Attachment of Primiparous Women: A Randomized Controlled Study. J Med Syst. 2023 Apr 1;47(1):44. doi: 10.1007/s10916-023-01942-3. PMID 37004692
- [Background] Ansari S, Abedi P, Hasanpoor S, Bani S. The Effect of Interventional Program on Breastfeeding Self-Efficacy and Duration of Exclusive Breastfeeding in Pregnant Women in Ahvaz, Iran. Int Sch Res Notices. 2014 Aug 19;2014:510793. doi: 10.1155/2014/510793. eCollection 2014. PMID 27379293
- [Background] Şenol DK, Pekyiğit AÇ. Effects of Breastfeeding Education Given in Childbirth Preparation Classes for Primipara Women on Their Perceived Prenatal Breastfeeding Self-Efficacy. Bozok Tıp Dergisi. 2021;11(2):15-21.
- [Background] Wells KJ, Thompson NJ, Kloeblen-Tarver AS. Development and psychometric testing of the prenatal breast-feeding self-efficacy scale. Am J Health Behav. 2006 Mar-Apr;30(2):177-87. doi: 10.5555/ajhb.2006.30.2.177. PMID 16533102
- [Background] Aydin A, Pasinlioglu T. Reliability and Validity of a Turkish version of the Prenatal Breastfeeding Self-Efficacy Scale. Midwifery. 2018 Sep;64:11-16. doi: 10.1016/j.midw.2018.05.007. Epub 2018 May 18. PMID 29852379
- [Background] Oras P, Ljungberg T, Hellstrom-Westas L, Funkquist EL. A breastfeeding support program changed breastfeeding patterns but did not affect the mothers' self-efficacy in breastfeeding at two months. Early Hum Dev. 2020 Dec;151:105242. doi: 10.1016/j.earlhumdev.2020.105242. Epub 2020 Oct 24. PMID 33137580
- [Background] 31. Bandura A. Self-efficacy. In. VS Ramachaudran. Encyclopedia of human behavior. 1994;4(4):71-81.
- [Background] Corby K, Kane D, Dayus D. Investigating Predictors of Prenatal Breastfeeding Self-Efficacy. Can J Nurs Res. 2021 Mar;53(1):56-63. doi: 10.1177/0844562119888363. Epub 2019 Nov 19. PMID 31744322
- [Background] Alyousefi N, Alemam A, Altwaijri D, Alarifi S, Alessa H. Predictors of Prenatal Breastfeeding Self-Efficacy in Expectant Mothers with Gestational Diabetes Mellitus. Int J Environ Res Public Health. 2022 Mar 30;19(7):4115. doi: 10.3390/ijerph19074115. PMID 35409796
- [Background] Ozdemir F, Yıkar SK, Nazik E. Predictors of breastfeeding self-efficacy in pregnant adolescents. Universa Medicina. 2022;41(3):254-62. https://doi.org/10.18051/UnivMed.2022.v41.254-262
- [Background] Başgöl Ş, Küçükkaya B. The Effect of Perceived Social Support on Prenatal Breastfeeding Self-Efficacy in Pregnants in Turkey: A web-based cross-sectional study. Kadın Sağlığı Hemşireliği Dergisi. 2022;8(3):133-43.
- [Background] Robinson KM, VandeVusse L. African American women's infant feeding choices: prenatal breast-feeding self-efficacy and narratives from a black feminist perspective. J Perinat Neonatal Nurs. 2011 Oct-Dec;25(4):320-8; quiz 329-30. doi: 10.1097/JPN.0b013e31821072fb. PMID 22071615
- [Background] Brockway M, Benzies K, Hayden KA. Interventions to Improve Breastfeeding Self-Efficacy and Resultant Breastfeeding Rates: A Systematic Review and Meta-Analysis. J Hum Lact. 2017 Aug;33(3):486-499. doi: 10.1177/0890334417707957. Epub 2017 Jun 23. PMID 28644764
- [Background] Khresheh RM, Ahmad NM. Breastfeeding self efficacy among pregnant women in Saudi Arabia. Saudi Med J. 2018 Nov;39(11):1116-1122. doi: 10.15537/smj.2018.11.23437. PMID 30397711
- [Background] Araban M, Karimian Z, Karimian Kakolaki Z, McQueen KA, Dennis CL. Randomized Controlled Trial of a Prenatal Breastfeeding Self-Efficacy Intervention in Primiparous Women in Iran. J Obstet Gynecol Neonatal Nurs. 2018 Mar;47(2):173-183. doi: 10.1016/j.jogn.2018.01.005. Epub 2018 Feb 3. PMID 29406289
- [Background] Feinstein J, Slora EJ, Bernstein HH. Telehealth can promote breastfeeding during the COVID-19 pandemic. NEJM Catalyst Innovations in Care Delivery. 2021;2(2). https://doi.org/10.1089/jwh.2021.0504
- [Derived] Metin A, Baltaci N. The effects of video-assisted breastfeeding education given to primiparous pregnant women on breastfeeding self-efficacy: randomized control study. BMC Pregnancy Childbirth. 2024 Feb 17;24(1):142. doi: 10.1186/s12884-024-06317-1. PMID 38368316
- See also: Türkiye Nüfus ve Sağlık Araştırması: Hacettepe Üniversitesi Nüfus Etütleri Enstitüsü; 2018. — https://fs.hacettepe.edu.tr/hips/dosyalar/Ara%C5%9Ft%C4%B1rmalar%20-%20raporlar/2018%20TNSA/2018_TNSA_Ozet_Rapor.pdf

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT06121973/Prot_SAP_ICF_000.pdf